CLINICAL TRIAL: NCT00977756
Title: IMPAACT P1058A: Intensive Pharmacokinetic Studies of New Classes of Antiretroviral Drug Combinations in Children, Adolescents and Young Adults
Brief Title: IMPAACT P1058A: Pharmacokinetic Effects of New Antiretroviral Drugs on Children, Adolescents and Young Adults
Status: Completed | Type: Observational
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: IMPAACT P1058A; U01AI068632 (NIH)
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: HIV Infections
Keywords: Treatment; Children; Integrase Inhibitors; Entry Inhibitors; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Atazanavir Sulfate; Ritonavir; Tenofovir; etravirine; Darunavir; Maraviroc; Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (11):
- Group G: Participants will receive a medication regimen including RAL + ATV + RTV.
  Interventions: Drug: Raltegravir (RAL); Drug: Atazanavir (ATV); Drug: Ritonavir (RTV)
- Group H: Participants will receive a medication regimen including RAL + TDF.
  Interventions: Drug: Raltegravir (RAL); Drug: Tenofovir (TDF)
- Group I: Participants will receive a medication regimen including ETV + DRV + RTV.
  Interventions: Drug: Ritonavir (RTV); Drug: Etravirine (ETV); Drug: Darunavir (DRV)
- Group J: Participants will receive a medication regimen including MVC + ATV + RTV.
  Interventions: Drug: Atazanavir (ATV); Drug: Ritonavir (RTV); Drug: Maraviroc (MVC)
- Group K: Participants will receive a medication regimen including MVC + LPV + RTV.
  Interventions: Drug: Ritonavir (RTV); Drug: Maraviroc (MVC); Drug: Lopinavir/ritonavir (LPV/r)
- Group L: Participants will receive a medication regimen including MVC + RAL + ETV.
  Interventions: Drug: Raltegravir (RAL); Drug: Etravirine (ETV); Drug: Maraviroc (MVC)
- Arm M: Participants will receive a medication regimen of DRV
- Arm N: Participants will receive a medication regimen of DRV
- Arm O: Participants will receive a medication regimen of unboosted ATV
- Arm P: Participants will receive a medication regimen of RPV
- Arm Q: Participants will receive a medication regimen of RPV

INTERVENTIONS:
Drug: Raltegravir (RAL) — 400 mg twice daily (BID)
  Other Names: Isentress
  Groups: Group G; Group H; Group L
Drug: Atazanavir (ATV) — 300 mg daily
  Other Names: Reyataz
  Groups: Group G; Group J
Drug: Ritonavir (RTV) — 100 mg daily, dosing by weight in Group I
  Other Names: Norvir
  Groups: Group G; Group I; Group J; Group K
Drug: Tenofovir (TDF) — 300 mg daily
  Other Names: Viread
  Groups: Group H
Drug: Etravirine (ETV) — 200 mg BID
  Other Names: Intelence
  Groups: Group I; Group L
Drug: Darunavir (DRV) — Dosing by weight
  Other Names: Prezista
  Groups: Group I
Drug: Maraviroc (MVC) — 150 mg BID in groups J and K; 600 mg BID in group L
  Other Names: Selzentry
  Groups: Group J; Group K; Group L
Drug: Lopinavir/ritonavir (LPV/r) — Coformulation of 400 mg lopinavir and 100 mg ritonavir, taken twice daily
  Other Names: Kaletra
  Groups: Group K

SUMMARY:
This study will examine drug and body interactions in children receiving anti-HIV treatment regimens using new medications. Drug regimens to be examined will feature the medications raltegravir (RAL), maraviroc (MVC), and etravirine (ETV). These drugs will not be provided through the study.

DETAILED DESCRIPTION:
Antiretroviral (ARV) medication regimens for children, adolescents and young adults are often prescribed based on drug resistance because of previous treatment history. In order to find an effective regimen, clinicians must often turn to newer drugs before they have been fully tested in adolescent or pediatric clinical trials. One of the first steps in testing these drugs is to assess the drug pharmacokinetics (PK), or interaction between drugs and body. This study, a follow-on protocol to the International Maternal Pediatric Adolescent AIDS Clinical Trials Group (IMPAACT) P1058 study, will test children, adolescents and young adults who have already been prescribed treatment regimens with new drugs. The study will examine the PK of medication combinations featuring raltegravir, a new drug in the new ARV class of entry inhibitors (EIs); maraviroc, a new drug in the new class of fusion inhibitors (FIs); and etravirine, a new drug in the class of non-nucleoside reverse transcriptase inhibitors (NNRTIs). Older medications may also be used to complete these regimens.

Participation in this study will last between 1 and 7 weeks and involve at least two clinic visits. The first is a screening and entry visit at which a medical history will be taken and a physical exam and blood test will be completed. The second visit will measure PK of the medications. During this visit, participants will complete the same measures as before-medical history, physical exam, blood test-and then be given a dose of their anti-HIV medication regimen. After receiving the medications, participants will be monitored and give blood samples after 1, 2, 4, 6, 8, and 12 hours. For Groups G, H, I, J, K and L an intensive 12-hour PK study will be scheduled after at least 30 days on the combination of interest. For all Groups, the intensive 12-hour PK study should be performed within 35 days (5 weeks) of screening/entry evaluations. Medications will not be provided through this study.

Results of the 12-hour medication monitoring tests will be delivered to participants' physicians within 6 weeks. If, based on these results, a physician decides to change the dosage of a participant's medication, that participant may be asked to complete a second PK visit. Participants must have received the revised dose for at least 14 days before the PK study can be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Certain laboratory values received within 5 weeks of the date of the screening or entry evaluations
* HIV infected
* Stable on the specified antiretroviral (ARV) regimen for 30 days prior to screening and entry. ARVs will not be provided through this protocol.
* Prescribed one of the regimens described in the study details by clinician on the basis of clinical need (although the availability of drug levels may have been a factor in clinical decision-making). The decision to initiate the regimen must have been solely that of the prescribing physician.
* On the ARV combination of interest for at least 14 days and within 5 weeks (35 days) of the date of screening results
* Body surface area (BSA) of at least 0.85 m2
* Participants in P1058 Version 1.0 and Version 2.0 who have switched to a regimen specified in the entry criteria are eligible for P1058A.
* Any licensed formulation that achieves these dosages, but without including a disallowed drug, may be used.
* Participants who have enrolled in P1058A (Groups G-L) and who subsequently switch to a different regimen specified in the entry criteria are eligible to re-register to a subsequent step of P1058A (re-consent required)
* Females must agree to use two reliable methods of contraception, one of which must be a barrier method, while taking study medications and for 6 weeks after study testing
* Documentation of presence of an R5-tropic virus at the start of treatment with maraviroc (MVC)

Exclusion Criteria:

* Pregnant or breastfeeding
* Hemoglobin level less than 8.5 g/dL
* Clinical evidence of pancreatitis as defined by moderate clinical symptoms
* Treatment with any anti-HIV or non-ARV drug that could interact with drugs under pharmacokinetic (PK) study in the 14 days prior to study entry
* Known allergy, sensitivity, or hypersensitivity to components of two or more study-specified drugs or their formulation

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: HIV infected children, adolescents and young adults who are receiving a regimen of antiretroviral drugs prescribed by their physician that includes one of the target combinations.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2002-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Steady state pharmacokinetics (PK) of raltegravir administered in combination with atazanavir/ritonavir or tenofovir or maraviroc/etravirine to older children, adolescents and young adults | Measured at baseline and 1, 2, 4, 6, 8, and 12 hours after dosing
Steady state PK of etravirine administered to older children, adolescents and young adults | Measured at baseline and 1, 2, 4, 6, 8, and 12 hours after dosing
Steady state PK of maraviroc administered in combination with atazanavir/ritonavir or lopinavir/ritonavir to older children, adolescents and young adults | Measured at baseline and 1, 2, 4, 6, 8, and 12 hours after dosing
Steady state PK of maraviroc (600 mg twice daily [BID]) given in combination with raltegravir and etravirine (a protease inhibitor [PI]-sparing regimen) to older children, adolescents and young adults | Measured at baseline and 1, 2, 4, 6, 8, and 12 hours after dosing

SECONDARY OUTCOMES:
Relationship between Tanner stage and the PK of the regimens of interest in children and adolescents | Measured at baseline and 1, 2, 4, 6, 8, and 12 hours after dosing
Relationships between the PK parameters and polymorphisms that may affect the antiretrovirals (ARVs) of interest in older children, adolescents and young adults | Measured at baseline and 1, 2, 4, 6, 8, and 12 hours after dosing
Adverse events associated with the ARVs of interest | Measured throughout
Steady state PK of darunavir/ritonavir administered to older children, adolescents and young adults | Measured at baseline and 1, 2, 4, 6, 8, and 12 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R. King, PharmD, Study Chair — University of Alabama at Birmingham; Ram Yogev, MD, Study Chair — Northwestern University Feinberg School of Medicine
Locations (35):
- United States (33):
  - Univ. of Alabama Birmingham NICHD CRS (5096), Birmingham, Alabama
  - Miller Children's Hospital Long Beach, CA NICHD CRS (5093), Long Beach, California
  - Usc La Nichd Crs (5048), Los Angeles, California
  - UCSD Mother, Child & Adolescent HIV Program(4601), San Diego, California
  - Univ. of California San Francisco NICHD CRS (5091), San Francisco, California
  - Harbor (UCLA) Medical Center NICHD CRS (5045), Torrance, California
  - Harbor Univeristy of California, Los Angeles (UCLA) Medical Center (603), Torrance, California
  - Childrens Hospital (U. Colorado, Denver) NICHD CRS (5052), Denver, Colorado
  - Children's National Medical Center (5015), Washington D.C., District of Columbia
  - South Florida CDC Ft Lauderdale NICHD CRS (5055), Fort Lauderdale, Florida
  - University of Miami Pediatric Perinatal HIV/AIDS CRS (4201), Miami, Florida
  - University of South Florida Tampa (5018), Tampa, Florida
  - Rush University Cook County (5083), Chicago, Illinois
  - Chicago Children's CRS (4001), Chicago, Illinois
  - University of Maryland NICHD CRS (5094), Baltimore, Maryland
  - Johns Hopkins University NICHD CRS (5092), Baltimore, Maryland
  - Children's Hospital of Boston NICHD CRS (5009), Boston, Massachusetts
  - Boston Medical Center Ped. HIV Program NICHD CRS (5011), Boston, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS (7301), Worcester, Massachusetts
  - New Jersey Medical School (NJ) (2802), Newark, New Jersey
  - New York University NY (5012), New York, New York
  - Metropolitan Hospital (5003), New York, New York
  - Columbia IMPAACT CRS (4101), New York, New York
  - SUNY Stony Brook NICHD CRS (5040), Stony Brook, New York
  - Bronx-Lebanon Hospital (6901), The Bronx, New York
  - Jacobi Medical Center Bronx (5013), The Bronx, New York
  - Duke University Medical Center (DUMC) (4701), Durham, North Carolina
  - The Children's Hosp. of Philadelphia IMPAACT CRS (6701), Philadelphia, Pennsylvania
  - St. Jude/UTHSC CRS (6501), Memphis, Tennessee
  - Texas Children's Hosp. CRS (3801), Houston, Texas
  - Harborview Medical Center NICHD CRS (5027), Seattle, Washington
  - Univ of Washington Children's Hospital Seattle (5017), Seattle, Washington
  - University of Washington NICHD CRS (5029), Seattle, Washington
- Puerto Rico (2):
  - San Juan City Hosp. PR NICHD CRS (5031), San Juan
  - University of Puerto Rico Pediatric HIV/AIDS Research (6601), San Juan

REFERENCES:
- [Background] Guidelines for the use of antiretroviral agents in pediatric HIV infection. Center for Disease Control and Prevention. MMWR Recomm Rep. 1998 Apr 17;47(RR-4):1-43. PMID 9572665
- [Background] Iwamoto M, Wenning LA, Petry AS, Laethem M, De Smet M, Kost JT, Breidinger SA, Mangin EC, Azrolan N, Greenberg HE, Haazen W, Stone JA, Gottesdiener KM, Wagner JA. Minimal effects of ritonavir and efavirenz on the pharmacokinetics of raltegravir. Antimicrob Agents Chemother. 2008 Dec;52(12):4338-43. doi: 10.1128/AAC.01543-07. Epub 2008 Oct 6. PMID 18838589
- [Background] Wenning LA, Friedman EJ, Kost JT, Breidinger SA, Stek JE, Lasseter KC, Gottesdiener KM, Chen J, Teppler H, Wagner JA, Stone JA, Iwamoto M. Lack of a significant drug interaction between raltegravir and tenofovir. Antimicrob Agents Chemother. 2008 Sep;52(9):3253-8. doi: 10.1128/AAC.00005-08. Epub 2008 Jul 14. PMID 18625763
- [Derived] Cressey TR, Hazra R, Wiznia A, Foca M, Jean-Philippe P, Graham B, King JR, Britto P, Carey VJ, Acosta EP, Yogev R; IMPAACT P1058A Team. Pharmacokinetics of Unboosted Atazanavir in Treatment-experienced HIV-infected Children, Adolescents and Young Adults. Pediatr Infect Dis J. 2016 Dec;35(12):1333-1335. doi: 10.1097/INF.0000000000001320. PMID 27583590